CLINICAL TRIAL: NCT03599960
Title: Combination Chemotherapy (Methotrexate, L-asparaginase, Idarubicin and Dexamethasone) in Patients With Newly Diagnosed Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Brief Title: Combination Chemotherapy in Patients With Newly Diagnosed BPDCN
Acronym: LpDessai
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: UMR1098, EFS BFC, BESANCON (Unknown); Centre Henri Becquerel (Other); Maisonneuve-Rosemont Hospital (Other); Centre Hospitalier Universitaire Dijon (Other); Inserm CIC1431, CHU Besancon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LpDessai
Record Dates: First submitted 2018-02-09; First posted 2018-07-26 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: All patients will receive 3 cycles of a combination of chemotherapy (Met/Ida/L-Asp/Dex)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — * Idarubicin 12mg/m2 IV at D1
  * Methotrexate at D1 (24H infusion, alkaline hydration, leucovorin rescue):
    * Patients <65y and albuminemia >35 g/l and CrCl (MDRD)>60 ml/min: 3000 mg/m²
    * Patients <65y and albuminemia <35 g/l and/or CrCl (MDRD) <60 ml/min: 1000 mg/m² IV
    * Patients ≥65y and albuminemia >35 g/l and CrCl (MDRD) > 60 ml/min : 1000 mg/m²
    * Patients ≥ 65y and albuminemia < 35 g/l and/or CrCl (MDRD) < 60 ml/min : 500 mg/m²
  * L-asparaginase (SPECTRILA) : 5000 units/m² IV at D2, 5, 8, 11 (switch to Erwinia asparaginase/Cirsantaspase 25 000 U/m² with the same drug regimen in case of hypersensitivity reactions or significant diminution of asparaginase activity)
  * Dexamethasone 40mg PO or IV at D1-4 (dose diminution at 20 mg for Age ≥65y)

SUMMARY:
Patients with suspected BPDCN and meeting eligibility criteria will be enrolled in the study. First, BPDCN diagnosis will be confirmed by anatomic pathology (Dr Petrella T, Montreal) and cytologic plus immunophenotyping analysis (Pr Garnache Ottou F, UMR1098 BESANCON). Patients will then receive three 21 days cycles of a combination of chemotherapy (Ida/Metho/L-asp/Dex), followed by an evaluation. Patients with complete response (CR) or complete response with incomplete bone marrow recovery (CRi) will undergo an allo- or auto-SCT and those who are not eligible to the transplantation will have successive 28 days cycles of chemotherapy (Metho/L-asp/Dex). Patients who did not respond to the treatment will be treated by physicians. All patients will be followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed BPDCN established by a blood or bone marrow immunophenotypic diagnosis by flow cytometric and/or by the anatomic pathology study of a skin biopsy using validated diagnostic criteria (Swerdlow SH CE et al., World Health Organisation Classification of Tumors, 2008; Garnache-Ottou et al., 2009; Angelot et al., 2012; Julia et al., 2014) or patients with confirmed isolated skin lesion.
* 18 years of age or older
* No prior cytotoxic therapy except <2 week of corticosteroids or hydroxyurea
* ECOG ≤2
* Written informed consent
* Affiliation to the French social security scheme

Exclusion Criteria:

* Cardiac contra-indication to anthracyclines: cardiac dysfunction events (NYHA grade 3 or 4 and/or LVEF<50%)
* Hepatocellular abnormalities except if considered related to the BPDCN:

  1. ASAT (SGOT) and/or ALAT (SGPT) > 5 x ULN
  2. Total bilirubin ≥ 2.5 x ULN
* Creatinine level >1.5x ULN or creatinine clearance (MDRD)<50 mL/mn
* Prior thrombotic event
* Active hepatitis B or C virus infection
* HIV positive
* Serious medical or psychiatric illness that could interfere with the completion of treatment
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Pregnant and lactating female patients
* Patients diagnosed with or treated for another malignancy within 2 years before study enrollment or with residual disease (basal cell carcinoma or cervical carcinoma in situ patients may be enrolled if they have undergone complete resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete response after 3 cycles of chemotherapy | 12 weeks (3 weeks after 3 cycles of chemotherapy (each cycle is 21 days))
  Proportion of patients with complete response after 3 cycles of chemotherapy

SECONDARY OUTCOMES:
Proportion of patients with response (complete or partial) after 3 cycles of chemotherapy | 12 weeks (3 weeks after 3 cycles of chemotherapy (each cycle is 21 days))
  Proportion of patients with response (complete or partial) after 3 cycles of chemotherapy
Overall survival | 24 months
  Overall survival
Relapse-free survival | 24 months
  Relapse-free survival
Residual L-asparaginase activity | 12 weeks (Day 8 of each chemotherapy cycle (each cycle is 21 days))
  Residual L-asparaginase activity
Anti-L-asparaginase antibodies levels | 12 weeks (Day 8 of each chemotherapy cycle (each cycle is 21 days))
  Evaluation of the titer of the anti-asparaginase antibody

OTHER OUTCOMES:
Minimal residual disease analysis | 24 months
  presence of PDC cell blast (CD56 +, NG2 +, BDCA2low, BDCA4low, CD123low, cTCL1high as measured by flow cytometry)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique de L'Europe, Amiens
  - Chu Besancon, Besançon

IPD SHARING:
Plan to Share IPD: No